CLINICAL TRIAL: NCT06666452
Title: The Feasibility Test of a COMbined Fatigue Intervention (COMFI) for People With Inflammatory Athritis
Brief Title: COMFI - a COMbined Fatigue Intervention
Acronym: COMFI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Center for Expertise in Rheumatology (Other)
Collaborators: Skaane University Hospital (Unknown); Odense Patient Data Explorative Network (Other); The Danish Rheumatism Association (Other); Region of Southern Denmark (Other); University of Southern Denmark (Other); Bristol Royal Infirmary (Unknown)
Responsible Party: Principal Investigator, Jette Primdahl, Professor in rheumatology rehabilitation, The Danish Center for Expertise in Rheumatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COMFI-Feasibility; S-20232000 - 110 (Other: The Scientific Regional Ethics Committees)
Record Dates: First submitted 2024-10-15; First posted 2024-10-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA); Spondyloarthritis (SpA); Inflammatory Arthritis
Keywords: Fatigue; Intervention; cognitive behavioural approach; Physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis; Arthritis; Fatigue; Motor Activity

STUDY DESIGN:
Masking Description: It is not possible to blind the intervention to the participants and the healthcare professionals in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The COMFI intervention
  Interventions: Behavioral: COMFI - a COMbined Fatigue Intervention

INTERVENTIONS:
Behavioral: COMFI - a COMbined Fatigue Intervention — The COMFI intervention is a 24-week group-based outpatient fatigue intervention consisting of 1) Six group sessions based on CBA covering topics such as fatigue and related factors, PA, trying out PA, energy management, and enhancing peer support 2) a seventh group session intended as a booster session in week 24, 3) one optional individual session in week 6-9 of the intervention, and 4) a support line in week 13-23 of COMFI.

SUMMARY:
Background: Inflammatory arthritis (IA) encompasses autoimmune rheumatic diseases, such as rheumatoid arthritis, psoriatic arthritis, and axial spondyloarthritis. Fatigue is highly prevalent in people with IA with 41-57% suffering from severe fatigue. Patients describe fatigue as overwhelming, unpredictable, challenging to manage, and affecting all areas of everyday life, including the ability to work. Studies have shown that interventions with physical activity or a cognitive behavioral approach can significantly reduce fatigue severity and/or impact in people with IA compared to usual care. To date, no studies have investigated the combined effect of CBA and PA on fatigue severity and impact in patients with IA. Therefore, the goal of this study is to test the feasibility of a newly developed fatigue intervention that combines a cognitive behavioral approach and physical activity (COMFI) in patients with inflammatory arthritis, who experience fatigue as a challenge in their everyday lives in Denmark and Sweden. The intervention will be tested in 4 groups (2 in Denmark and 2 in Sweden), and the participants will participate in 7 group sessions and 2 focusgroups interview in the evaluation.

The primary outcome for the participants is fatigue, measured through patient-reported outcomes at baseline, 3, 6, and 12 months after baseline.

This study will show if the intervention is feasible in practice and meaningful for the participants.

DETAILED DESCRIPTION:
Background: Inflammatory arthritis (IA) encompasses chronic autoimmune rheumatic diseases, such as rheumatoid arthritis (RA) and spondyloarthritis (which includes psoriatic arthritis, PsA, and axial spondyloarthritis, axSpA). In Denmark, the prevalence of people living with RA, PsA, or axSpA is approximately 50,000, 25,000, and 5,000 respectively. The characteristics of IA-related symptoms encompass swollen joints, stiffness, loss of physical function, pain, fatigue, sleep problems, and emotional distress. Despite advances in pharmacological treatment over the last decades and treat-to-target strategies aiming to reduce disease activity for people with IA, many still struggle with the substantial impact of fatigue on their everyday lives. Fatigue is highly prevalent in people with IA with 41-57% suffering from severe fatigue. The patients describe fatigue as overwhelming, unpredictable, disabling, challenging to manage, and affecting all areas of everyday life, including their health-related quality of life (HRQOL), performance of activities, and participation in daily living. Participation includes workability, which is important for a person's identity to be able to work, and it provides a sense of purpose and quality of life. Patients expressed the need for support to manage the impact of IA-related fatigue on everyday life. Besides the individual burden of living with fatigue, the high levels of absenteeism, and work disability contribute to societal and economic costs. Thus, from both a patient and a societal perspective, interventions aiming to reduce the impact of fatigue in people with IA are needed.

To encompass the complex and multidimensional nature of fatigue, a management approach incorporating pharmacological and non-pharmacological interventions is needed. Reviews on non-pharmacological interventions for fatigue in people with RA have shown that psychosocial and physical activity interventions can reduce fatigue severity. Additionally, studies have documented that interventions with physical activity or a cognitive behavioral approach significantly reduced fatigue severity and/or impact in people with IA compared to usual care. One of those, the Lessening the Impact of Fatigue in Inflammatory Rheumatic Disease Trial (LIFT) study compared three arms: 1) usual care 2) usual care and a cognitive behavioral approach, and 3) usual care and a personalized exercise program. Both a cognitive behavioral approach and a personalized exercise program, in addition to usual care, reduced fatigue severity and impact compared to usual care only. In the Reducing Arthritis Fatigue: clinical Teams using CB approaches (RAFT) study, a cognitive behavioral approach was delivered in a face-to-face group intervention by trained members of the rheumatology team in addition to usual care significantly reduced fatigue impact and increased self-efficacy compared to usual care only. Additionally, the study showed high patient satisfaction and attendance in the cognitive behavioral approach group. To include both a cognitive behavioral approach and a personalized exercise program may reduce the severity and impact of fatigue further, but to date, no studies have investigated the combined effect of a cognitive behavioral approach and physical activity on fatigue severity and impact in patients with IA.

Thus, the aim of this study is to evaluate the feasibility (acceptability, dose, and fidelity) and preliminary outcomes of the developed COMFI, which combines a cognitive behavioral approach and physical activity support for people with IA to improve the management of fatigue and to reduce fatigue severity and -impact among patients with IA in Soenderborg, Denmark and Lund, Sweden.

Methods The testing of COMFI will be guided by the UK Medical Research Council (MRC) framework for developing and evaluating Complex Interventions.

This feasibility study is a single-arm interventional study to assess the COMFI intervention, which is a newly developed 24-week group-based outpatient fatigue intervention consisting of 1) Six group sessions based on a cognitive behavioral approach covering topics such as fatigue and related factors, physical activity, trying out physical activity, energy management, and enhancing peer support 2) a seventh group session intended as a booster session in week 24, 3) one optional individual session in week 6-9 of COMFI, and 4) a support line in week 13-23 of COMFI. Additionally, the participants will participate in 2 focus group interviews after the sixth and seventh sessions to enable a qualitative evaluation of the intervention.

The groups in the intervention will consists of 8-10 participants, and the intervention will be tested in two groups in each site (four in total), which means 16-20 patients with IA from each of the involved hospitals will be included in this feasibility test.

Recruitment in Denmark: Before clinical consultations, the patient completes questionnaires in the Danish Rheumatology Quality Database (DANBIO), including. VAS fatigue. If VAS fatigue ≥60, a text appears on the screen with information about the project and the opportunity to add their phone number for further contact. The research department then contacts eligible patients to provide more information about the project and request written consent for participation and accessing medical records and data in DANBIO. Eligible patients receive written information and consent material electronically or via postal mail.

Recruitment in Sweden: Manually check in Swedish Rheumatology Quality Register (SRQ) for eligible patients and contact them to inquire if they are interested in participating in the project. The following procedure will be the same as in Denmark.

Data collection: Outcomes will be measured at baseline (week 0), end of intervention (week 12), after the booster session (week 24), and at follow-up (week 52). Patient-reported outcomes will be collected through the software program RedCap, and the databases DANBIO and SRQ. Physical measurements or tests will be imputed into REDCap. Additionally, Information on attendance, time use, etc. will be recorded by the health professionals in a "logbook".

Ethics The project is conducted in line with the Helsinki Declaration, and the Danish and Swedish codex for research. The project is registered at the Danish Data Protection Agency and the local regional scientific ethical committee in the Region of Southern Denmark declared that the project does not need formal approval (case number: S-20232000 - 110). Ethical approval from The Swedish Ethical Review Authority has been obtained. All participants will receive oral and written information about the study and provide written consent to participate. Data will be pseudo-anonymized and measures to protect the integrity of the participants will be taken. Data storage and management in Open Patient Data Explorative Network (OPEN) (a secure application in the Region of Southern Denmark), which is a secure application in the Region of Southern Denmark which complies with the European General Data Protection Regulation (GDPR) and Danish law for data protection.

ELIGIBILITY:
Inclusion Criteria:

1. Current fatigue level (VAS-Fatigue: The VAS-fatigue has to be 60 or above.
2. Must have experienced fatigue as a challenge for at least the last 3 months
3. A rheumatologist-confirmed diagnosis of Rheumatoid Arthritis, Psoriatic Arthritis, or Spondyloarthritis
4. The patient is in a stable phase regarding disease activity. This means no current plans to adjust pharmacological treatment, and no changes in treatment in the last 3 months (DMARDs or steroids) incl. steroid injections.
5. Must be affiliated with the Danish Hospital of Rheumatic Diseases or Skaane University Hospital in Lund.
6. Age ≥18 years.
7. Must be able to speak and write Danish or Swedish well enough to participate in group discussions without an interpreter.
8. The participant must be interested in actively participating and making changes to daily life to improve their condition.

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Critical/serious illness:

   * Diseases with an expected survival of < 2 years (e.g., cancer)
   * Heart failure with NYHA class 3 or 4
   * Kidney failure with eGFR < 30
   * Severe anemia - hemoglobin ≤ 5.0 mmol/L
3. Clarification of known diseases, which must be well-treated or in remission:

   * Diabetes: HbA1c >53 mmol/mol is excluded if dysregulated
   * Thyroid disease: TSH: 0.4-4.0 mE/L. Excluded if dysregulated
4. A medical condition that would make the proposed interventions unsuitable/impossible for group participation or hinder the ability to give informed consent:

   * Unstable psychiatric illness
   * Dementia or other severe cognitive problems
   * Hearing loss/use of hearing aids (it must be clarified how the person feels about being in a group setting)
   * Other physical or mental conditions with the above effect
5. Conditions that may be the primary cause of fatigue:

   * Long-term effects after COVID-19
   * Chronic fatigue syndrome
6. Participation in another research project that could affect fatigue (WORK-ON, INSELMA, SPINCODE)
7. Participation in the fatigue program for hospitalized patients or support in another way specifically related to fatigue
8. The participant must not have a planned rehabilitation stay (e.g., Danish Rheumatism Hospital, Sano, Montebello) or another program elsewhere that works with fatigue
9. If the participant cannot commit to attending on the scheduled dates in one of the two programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue - the Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF-MDQ) | At Baseline, and 3, 6, and 12-month follow-up
  Fatigue is measured through the Danish and Swedish versions of the questionnaire the Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF-MDQ). The BRAF-MDQ covers four subscales assessing physical fatigue, emotional fatigue, cognitive fatigue, and the impact of living with fatigue, which are scored individually and summed to reach a total fatigue score ranging from 0-70, with higher scores indicating more severe fatigue.
Fatigue - the Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales (BRAF-NRS v2) | At Baseline, and 3, 6, and 12-month follow-up
  Fatigue is measured through the Danish and Swedish versions of the questionnaire the Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales (BRAF-NRS v2) for fatigue level (severity), effect on life (impact), and coping. BRAF-NRS v2s three separate numerical rating scales are scored from 0-10, and for severity and impact 10 represents worse level or impact of fatigue, where for coping 10 is better at coping).

SECONDARY OUTCOMES:
Physical activity - objectively measured | Baseline and at 6-month follow-up
  Physical activity will be objectively measured through an accelerometer from SENS motion. The participants will wear an accelerometer for 7 days before starting the intervention and before participating in session 7.
Physical activity - Diary | Baseline and at 6-month follow-up
  The accelerometer will be combined with a diary tracking sleep, movement/work, and sedentary time to further qualify the results from the accelerometer.
Physical activity - Physical fitness test | Baseline
  Participants will perform the Aastrand bike sub-maximal physical fitness test (aerobic capacity).
Physical activity - Patient-reported | At Baseline, and 3, 6, and 12-month follow-up
  Physical activity will be measured through the questionnaire International Physical Activity Questionnaire (IPAQ), which enables the calculations of MET.
Health-related quality of life | At Baseline, and 3, 6, and 12-month follow-up
  European Quality of Life - 5 Dimensions (EQ-5D-5L) is a generic questionnaire to assess population health. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The EQ-5D-5L index ranges from 0.00 to 1.00. The higher the score, the better the health-related quality of life is.
Health-related quality of life visual analog scale (VAS) | At Baseline, and 3, 6, and 12-month follow-up
  European Quality of Life - 5 Dimensions VAS (EQ-5D-5L VAS) ranges from 0-100 with a higher score representing better health-related quality of life.
Mental Well-being | At Baseline, and 3, 6, and 12-month follow-up
  WHO-5 Well-being Index, The 5-item Well-Being Index is a generic rating scale measuring subjective well-being. WHO-5 ranges from 0-100, and a lower score reflects lower/less mental well-being.
Stress | At Baseline, and 3, 6, and 12-month follow-up
  Stress is measured through the questionnaire 10-Item Perceived Stress Scale (PSS-10), which assesses stress levels over the past four weeks. PSS-10 has sum scores ranging from 0 to 40. Higher scores reflect greater perceived stress.
Pain level | At Baseline, and 3, 6, and 12-month follow-up
  Pain is measured with the Visual analogue scale (VAS) pain, measuring self-rated pain at the moment from 0-10, a higher scores reflect worse pain.
Disease impact | At Baseline, and 3, 6, and 12-month follow-up
  Participants will assess the impact of the disease through the isual Analogue Scale (VAS) patient global impact of the disease. This scale ranges from 0 to 100, and higher scores reflect higher impact of disease.
Sleep | At Baseline, and 3, 6, and 12-month follow-up
  Sleep is measured through the questionnaire the Insomnia Severity Index (ISI). The scale ranges from 0-28. The higher the score, the more impaired sleep/worse sleep problems.
Physical function | Baseline
  Physical function is measured through the questionnaire the Multi-dimensional Health Assessment Questionnaire (MD-HAQ). MD-HAQ ranges from 0 to 3, and a higher score reflects a higher degree of physical limitations.

OTHER OUTCOMES:
Disease activity for patients with RA | Baseline
  The DAS28-CRP is a measure of disease activity in RA; assessing 28 specified joints, serum inflammatory markers, and a visual analog scale (0-10) of the patient's global function. A score greater than 5.1 indicates active disease and less than 3.2 indicates well-controlled disease.
Disease activity for patients with SpA and PsA | Baseline
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The scale ranges from 0-100. The higher the number, the more disease activity.
Supplementary question regarding sleep duration | At Baseline, and 3, 6 and 12 months follow-up
  In the past 4 weeks, how many hours and minutes did you sleep on an average weekday night?

CONTACTS AND LOCATIONS:
Overall Officials: Jette Primdahl, Professor, Study Director — The Danish Center for Expertise in Rheumatology
Locations (2):
- The Danish Hospital for Rheumatic Diseases, Sønderborg, Denmark, Denmark
- Skåne University Hospital, Lund, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No